CLINICAL TRIAL: NCT03970590
Title: Continuing the Conversation: A Multi-site RCT Using Narrative Communication to Support Hypertension Self-Management Among African-American Veterans
Brief Title: Continuing the Conversation: Using Narrative Communication to Support Hypertension Self-management in African American Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 17-185
Record Dates: First submitted 2019-05-30; First posted 2019-05-31 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Hypertension
Keywords: hypertension; Minority Health; health behavior; text messaging
MeSH Terms: conditions — Hypertension; Health Behavior

STUDY DESIGN:
Intervention Model Description: The investigators will conduct an RCT testing the CTC intervention (video viewing, selection of preferred narrative, narrative-aligned text messages) compared to assessment text messages alone.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CTC (Experimental): An integrated peer narrative-based intervention (VIEW > SELECT > GET), beginning with VIEW In-person viewing of VA Stories narratives, followed by SELECT a favorite Veteran Storyteller, and then GET favorite Storyteller "narrative-aligned" text messages over 6 months
  Interventions: Behavioral: CTC Intervention
- Control (Active Comparator): 6-month HTN management assessment text messages without narrative component
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: CTC Intervention — An integrated peer narrative-based intervention (VIEW > SELECT > GET), beginning with VIEW In-person viewing of VA Stories narratives, followed by SELECT a favorite Veteran] Storyteller, and then GET favorite Storyteller "narrative-aligned" text messages over 6 months
  Other Names: CTC
  Arms: CTC
Behavioral: Control — 6-month HTN management assessment text messages without narrative component
  Other Names: Active Comparator
  Arms: Control

SUMMARY:
In this study the investigators will conduct a randomized controlled trial aimed at improving hypertension self-management and lowering blood pressure (BP) in African-American Veterans. In this study, the investigators 'begin the conversation' by showing previously created videos to Veteran participants, inviting them to select the peer narrative that is most compelling. The investigators then 'continue the conversation', offering longitudinal support via 6 months of narrative-aligned text messages. Texts will cover key subject areas, providing education, reminders and periodic assessments, and include quotations derived from and aligned with transcripts from the chosen narrative. The investigators will measure the intervention's impact on BP, self-efficacy and self-management behaviors, and conduct a cost analysis.

DETAILED DESCRIPTION:
This project proposes to Continuing the Conversation, following a previous study in which the investigators used storytelling in African Americans Veterans, to create videos of how they manage their blood pressure. The investigators demonstrated significant differences in intention to change HTN management behavior immediately after video viewing; however, effects on blood pressure were not sustained, and six-month outcomes revealed only modest benefit over control (p = 0.06). The investigators' findings highlight the need for longitudinal support to sustain the storytelling effect. The proposed study provides longitudinal support via text messages, incorporating content from the participant's chosen peer narrative as a means of sustaining motivation and engagement in HTN self-management.

The proposal, "Continuing the Conversation," is a novel integration of peer narrative communication into technology. While use of an informatics tools (texting) as a channel to support self-management is not novel per se, the extension of a narrative via longitudinal texting is an innovative mechanism for supporting and sustaining HTN self-management behaviors. The investigators' Specific aims include:

Aim 1. Refine and Pilot the Continuing the Conversation (CTC) intervention. Previously, the investigators created video-recorded stories told by African-American Veterans with HTN, describing their self-management strategies. The investigators will refine CTC by adapting content from these videos to create narrative-aligned texts and will pilot CTC.

Aim 2. Test CTC by conducting a randomized controlled trial. CTC 'begins the conversation' by showing Veteran Story videos to participants, then inviting participants to select a preferred narrative. The investigators then 'continue the conversation,' offering longitudinal support via 6 months of narrative-aligned text messages. Messages cover key HTN content, providing education, reminders and weekly assessments, and include quotations derived from the chosen narrative. Control participants receive weekly assessment texts addressing the same key HTN self-management behaviors.

Aim 3. Evaluate CTC effectiveness, and mediating factors, and conduct a cost analysis. The investigators hypothesize that, for the CTC Intervention group as compared to the control: (H1)the difference in blood pressure from baseline to 6 months (primary outcome) will favor CTC intervention compared with the change in control. (H2): Self-efficacy and HTN management behaviors during 6-month follow-up will be greater for those in the CTC intervention group than control.

Methods: In a randomized controlled trial, 600 African-American Veterans with poorly controlled HTN will be recruited from 2 VA healthcare sites with known disparities in HTN control. The investigators will use within-site randomization (CTC vs. Control). Outcomes will include blood pressure, self-efficacy and HTN management behaviors. Longitudinal texts are designed to bring the storyteller back into the Veteran's everyday life, reminding and reinforcing as Veterans engage in the numerous daily decisions that will impact their blood pressure and their lives. Incorporating peer content into text messages in this way is highly innovative and offers a promising approach to supporting Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who have been receiving care at the recruiting VA site for 1 year prior to recruitment
* With 2 or more visits documented over the past year
* Veterans who have documented HTN (ICD10 diagnosis codes: I10-essential HTN) during this 1-year period
* Patients who self-identify as African American or Black
* Participants must be on at least one medication for BP
* Need to have access to their own or a family member's cell phone or smart phone for participation

  * Must be willing to use this phone for receipt of text messages over a 6-month period

Exclusion Criteria:

* Veterans who participated in our previous VA Stories study
* Veteran who fail the memory and concentration questions asked in the screening survey
* Pregnant Veterans (verified by self-report)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Cutrona, MD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (3):
- United States (3):
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to report on our primary outcome. In addition, during and following this trial, the investigators will provide materials to our operational partner, the Office of Connected Care (OCC), for presentations to National Leadership Council including to VISN Directors and also explore other avenues for dissemination.

REFERENCES:
- [Result] DeLaughter KL, Fix GM, McDannold SE, Pope C, Bokhour BG, Shimada SL, Calloway R, Gordon HS, Long JA, Miano DA, Cutrona SL. Incorporating African American Veterans' Success Stories for Hypertension Management: Developing a Behavioral Support Texting Protocol. JMIR Res Protoc. 2021 Dec 1;10(12):e29423. doi: 10.2196/29423. PMID 34855617
- [Derived] Cutrona SL, McDannold SE, DeLaughter KL, Fix GM, Shimada SL, Bokhour BG, Gordon HS, Pope C, Smith BM, Ndiwane N, Gardner J, DeFelice DC, Bal ES, Long JA. Text Messaging and Video Stories to Support Hypertension Self-Management in Black Veterans: A Randomized Clinical Trial. JAMA Netw Open. 2025 Nov 3;8(11):e2541342. doi: 10.1001/jamanetworkopen.2025.41342. PMID 41191358

RESULTS

PARTICIPANT FLOW:
Groups:
- CTC Intervention: An integrated peer narrative-based intervention (VIEW > SELECT > GET), beginning with VIEW In-person viewing of VA Stories narratives, followed by SELECT a favorite Veteran Storyteller, and then GET favorite Storyteller "narrative-aligned" text messages over 6 months
Period: Overall Study
Arm/Group | CTC Intervention | Control
Started | 300 | 300
Completed | 289 | 262
Not Completed | 11 | 38

BASELINE CHARACTERISTICS:
Population: Participant recruitment goals were met at 300 enrolled for each of the two study sites. Randomized assignment to Intervention/Control was used, resulting in 300 participants for each arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | CTC Intervention | Control | Total
Number analyzed (Participants) | 300 | 300 | 600
Age, Categorical [Count of Participants; unit: Participants] — Population: Some participants declined to answer certain questions.
  Participants
    number analyzed (Participants) | 288 | 298 | 586
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 148 | 150 | 298
    >=65 years | 140 | 148 | 288
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Some participants declined to answer.
  years
    number analyzed (Participants) | 288 | 298 | 586
    (all) | 64 (9) | 64 (9) | 64 (9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Some participants declined to answer.
  Participants
    number analyzed (Participants) | 299 | 298 | 597
    Female | 70 | 58 | 128
    Male | 229 | 240 | 469
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 300 | 300 | 600
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 300 | 300 | 600

OUTCOME MEASURES:

1. Primary Outcome: BP Measurement Change at Follow-up
Description: Blood Pressure (H1), will be calculated / performed to detect a difference in the change in both Diastolic and Systolic BP, comparing intervention and control.
Time Frame: From enrollment to the time of follow-up, up to 8 months
Population: Participants who completed study follow-up.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CTC Intervention | Control
Number analyzed (Participants) | 262 | 264
mmHg
  Systolic | 132 (17) | 133 (15)
  Diastolic | 80 (11) | 78 (12)

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected during the study period from enrollment to the time of follow-up, up to 8 months for each participant, and more specifically, at the time of follow-up if study staff learned of a participant death. Participants were enrolled beginning January 2021, and follow-ups were conducted beginning July 2021. Adverse event data collection was completed May 4, 2023, at study completion.
Arm/Group | CTC Intervention | Control
All-Cause Mortality (participants affected / at risk) | 5/300 | 4/300
Serious Adverse Events (participants affected / at risk) | 0/300 | 0/300
Other Adverse Events (participants affected / at risk) | 0/300 | 0/300

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT03970590/Prot_001.pdf
  • Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT03970590/SAP_002.pdf
  • Informed Consent Form (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT03970590/ICF_000.pdf